CLINICAL TRIAL: NCT04073758
Title: Comparing Analgesic Requirements in Patients Receiving Nuss Operation Using Remifentanil or Dexmedetomidine as Anesthetic Adjuvants
Brief Title: Comparison of Analgesic Requirements in Patients Receiving Nuss Operation Using 2 Different Anesthetic Adjuvants
Acronym: ARNRD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jung Min Koo (Other)
Responsible Party: Sponsor-Investigator, Jung Min Koo, Principal Investigator, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KC19MCSI0334
Record Dates: First submitted 2019-08-20; First posted 2019-08-29 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Chest Wall Disorder
Keywords: Pectus Excavatum
MeSH Terms: conditions — Funnel Chest | interventions — Dexmedetomidine; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remifentanil group (Sham Comparator): In both interventional groups, Sevoflurane is used as an inhalational agent, in 0.5-1.5% age-adjusted Minimal Alveolar Concentration (MAC). As explained above, remifentanil is infused with Target Controlled Infusion pump, and concentration is adjusted so that Bispectral index (BIS) is maintained as 40-60, which means that the patients are maintained in general anesthesia. Remifentanil is usually infused with the effect site concentration of 2.0 to 6.0 ng/ml during general anesthesia. If bradycardia or hypotension develops due to remifentanil infusion, the infusion rate could be reduced, or inotropic, vasopressor, anticholinergic agents can be used (ephedrine, atropine, etc.) to correct the side effects of the drug, or the drug infusion can even be ceased. At the end of the surgery when skin closure starts, remifentanil infusion will be stopped.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine group (Active Comparator): In both interventional groups, Sevoflurane is used as an inhalational agent, in 0.5-1.5% age-adjusted MAC (Minimal Alveolar Concentration). As explained above, dexmedetomidine is infused with syringe pump, and concentration is adjusted so that Bispectral index (BIS) is maintained as 40-60, which means that the patients are maintained in general anesthesia. Dexmedetomidine is loaded for 10 minutes in 1mcg/kg, and then infusion rate is set between 0.4 to 0.6mcg/kg/hour for this study. If bradycardia or hypotension develops due to remifentanil infusion, the infusion rate could be reduced, or inotropic, vasopressor, anticholinergic agents can be used (ephedrine, atropine, etc.) to correct the side effects of the drug, or the drug infusion can even be ceased. At the end of the surgery when skin closure starts, dexmedetomidine infusion will be stopped.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Comparing effects of remifentanil versus dexmedetomidine
  Other Names: Remifentanil

SUMMARY:
Nowadays, general anaesthesia is carried under "balanced anesthesia technique" in which many anesthetic adjuvants are used simultaneously, including opioid analgesics in order to reduce the amount of inhalation agents. The most popular adjuvants used are remifentanil, which is an opioid analgesic, and dexmedetomidine. Both of these agents are short acting, can be infused with targeted concentrations, excreted shortly from the body with stable hemodynamics.

Remifentanil, when infused for more than 2 hours, causes hyperalgesia to increase the amount of pain postoperatively as well as the amount of opioid analgesics. However, dexmedetomidine does not cause hyperalgesia and is known to have an opioid -sparing effect. In our center.

In this study, we aim to compare the effects of remifentanil and dexmedetomidine on postoperative pain in patients undergoing Nuss procedure, which is a very painful operation on the chest wall.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged >20
2. Patients undergoing Nuss bar operation (pectus excavatum repair surgery)
3. American Society of Anesthesiologists classification I ~ III

Exclusion Criteria:

1. Drug abuse history
2. Chronic pain in need of continuous opioid analgesics administration
3. History of psychiatric diseases
4. Preoperative bradycardia (heart rate < 50/min) or arrythmia
5. Cardiac diseases other than diabetes or hypertension - coronary artery disease, ischemic heart disease
6. Moderate liver or kidney dysfunction
7. Pregnant or breast feeding women
8. Hypersensitivity to the study drugs
9. Patients who do not agree to participate

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-09-02 (Actual); Primary Completion 2021-02-21 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | Between 1~6 hours postoperatively.
  Pain scale ranges from 0 to 10. 0 means no pain at all, and 10 being the most severe pain anyone can imagine.
Visual Analogue Scale | Between 6~12 hours postoperatively.
  Pain scale ranges from 0 to 10. 0 means no pain at all, and 10 being the most severe pain anyone can imagine.
Visual Analogue Scale | Between 12~24 hours postoperatively.
  Pain scale ranges from 0 to 10. 0 means no pain at all, and 10 being the most severe pain anyone can imagine.
Visual Analogue Scale | Between 24~48 hours postoperatively.
  Pain scale ranges from 0 to 10. 0 means no pain at all, and 10 being the most severe pain anyone can imagine.

SECONDARY OUTCOMES:
Amount of postoperative intravenous patient controlled analgesics (PCA) used | At 60 minutes after the end of surgery
Amount of fentanyl used postoperatively at the recovery unit | At 60 minutes after the end of surgery
  Amount in micgrograms per wegith in kilograms (migrogram/kilogram)
Time needed for postoperative rescue opioid analgesics | At 60 minutes after the end of surgery
Amount of remifentanil or dexmedetomidine used intraoperatively | Immediately at the end of the surgery
Intraoperative hemodynamic change: Systolic blood pressure | 1 minute after monitoring (of blood pressure, heart rate, pulse oxymeter and electrocardiogram) starts, when the patient arrives at the operating room
Intraoperative hemodynamic change: Diastolic blood pressure | 1 minute after monitoring (of blood pressure, heart rate, pulse oxymeter and electrocardiogram) starts, when the patient arrives at the operating room
Intraoperative hemodynamic change: mean blood pressure | 1 minute after monitoring (of blood pressure, heart rate, pulse oxymeter and electrocardiogram) starts, when the patient arrives at the operating room
Intraoperative hemodynamic change: heart rate | 30 minutes after the induction of anesthesia
Intraoperative hemodynamic change: mean blood pressure | At the end of the surgery, average of 90minutes after the induction of anesthesia
Intraoperative hemodynamic change: heart rate | At the end of the surgery, average of 90minutes after the induction of anesthesia
Intraoperative hemodynamic change: Systolic blood pressure | At the end of the surgery, average of 90minutes after the induction of anesthesia
Intraoperative hemodynamic change: Diastolic blood pressure | At the end of the surgery, average of 90minutes after the induction of anesthesia
Rescue drugs (inotropics or vasopressors) used in order to correct hypotension or bradycardia | Intraoperatively
Postoperative complications | Between 1~6 hours postoperatively
  Number of events that happened to the patient: e.g. Yes or No, and how many times. Nausea/vomiting, hypotension, respiratory depression, urinary retension, dizziness, transient cease in use of intravenous patient controlled analgesics (PCA)
Postoperative complications | Between 12~24 hours postoperatively
  Number of events that happened to the patient: e.g. Yes or No, and how many times. Nausea/vomiting, hypotension, respiratory depression, urinary retension, dizziness, transient cease in use of intravenous patient controlled analgesics (PCA)
Postoperative complications | Between 24~48 hours postoperatively
  Number of events that happened to the patient: e.g. Yes or No, and how many times. Nausea/vomiting, hypotension, respiratory depression, urinary retension, dizziness, transient cease in use of intravenous patient controlled analgesics (PCA)

CONTACTS AND LOCATIONS:
Overall Officials: Jung Min Koo, M.D, Principal Investigator — Data recruitment
Locations (1):
- Jung Min Koo, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No